CLINICAL TRIAL: NCT02201836
Title: The Effects of Music Therapy as a Complementary Intervention in the Treatment of Pediatric Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 142-04
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- One time music therapy session (Active Comparator): One time music therapy session which consists of music meditation, including as assessment/evaluation of confined body breathing function as expressed through drawing and coloring post music imagery session. This is followed by an entrainment wind playing/breath expansion music therapy intervention. At the end of the session, the subjects are given a donated wind instrument for play at home.
  Interventions: Other: One time music therapy
- Weekly group music therapy intervention (Active Comparator): The weekly group music therapy intervention consists of children and teens using guided visualization and expressing their fears and or fantasies related to breathing with one another. This is followed by creative music improvisations with part-playing on flutes, slide whistles, recorders and melodicas.
  Interventions: Other: Group music therapy
- Control (No Intervention)

INTERVENTIONS:
Other: One time music therapy
  Arms: One time music therapy session
Other: Group music therapy
  Arms: Weekly group music therapy intervention

SUMMARY:
The onset of asthma is particularly frightening for children. When the symptoms of asthma decrease, children and parents forget about the maintenance and control of breath and lung volume. Because adherence is so poor, asthma is known as the emergency room illness. The playing of a wind instrument is a unique way to provide a creative means for children and teens to understand both the impact of diaphramatic breathing and their ability to control it as well. This study builds upon the evidence, though sparse, that suggest that the blowing of a wind instrument with clinical music therapy intervention strengthens the muscles of breathing and fortifies the incentive toward attending to the daily symptoms and general management of asthma.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 7 and 18
* diagnosed with asthma

Exclusion Criteria:

* over 18

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2006-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 6 months
  The Juniper Questionnaire is a stringent quality of life measure that provides interview for children and teens and their parents. It is one of the few scales that requires these interviews to occur separately, so that children and parents do not feel compelled to answer what they think the other desires to hear. We also used take home journals and a comprehensive medical assessment to learn of ER visits, missed school days, avoidance of medication, and allergens in the home, as well as socio-economic status - these factors are known in the literature to effect outcomes and exacerbations with this population.

SECONDARY OUTCOMES:
Increase volume capacity | 6 months
  Spirometry enabled us to analyze the possible effects of wind playing on the child's breathing

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Loewy, DA, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States